CLINICAL TRIAL: NCT05213962
Title: Prospective Observational Study for Local Radiotherapy in Breast Cancer Patients Receiving Nipple Sparing Mastectomy With Breast Reconstruction
Brief Title: Local and Regional Radiotherapy for Nipple Sparing Mastectomy With Implant
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal Investigator, National Cancer Center, Korea
Other Study IDs: NCC2021-0335
Record Dates: First submitted 2021-12-21; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prospective observational study of radiation therapy is conducted on the nipple-areola complex(close resection margin at primary tumor site) or regional lymph nodes(including axilla and supraclavicular lymph node) with a high risk of local recurrence in nipple-sparing mastectomy with reconstruction, we're going to analysis the effects of radiation therapy and cosmetic effects.

By evaluating survival rate, recurrence pattern(local lymph node and metastasis to the whole body), side effects, cosmetic effects, from the patients who have gone through Nipple Sparing Mastectomy with reconstruction.

DETAILED DESCRIPTION:
For the last 20years, Breast Conservation Surgery and postoperative radiotherapy were the well established standard treatment, proven by various clinical trial studies, About 20-50% of breast cancer patients with large tumors, small breasts, or multiple tumors were still considered for Radical mastectomy.

In this case, Nipple Areola Complex (NAC) removal, significantly increases the amputation sensation of the patient and reduces breast contour, cosmetic satisfaction, physical balance, and psychological burden.

For this reason, recently, Nipple Sparing Mastectomy with reconstruction, which does not reduce treatment effect and maintain breast contour function is more considered.

It is reported that from Radical mastectomy specimens, possible tumor cell invasion in Nipple-Areola Complex is about 20%(0-58%).

local recurrence of breast cancer patient for nipple sparing mastectomy is reported to be about 0-28.4%.

Also, while operating a conserved Nipple Areola Complex (NAC) specimen, the false-negative rate of frozen section examination is 1.5-9.3%.

Therefore, due to the limitations of these pathological examinations, the possibility of residual tumor cells in the Nipple-Areola Complex cannot be excluded because that is unidentified and preserved in the tumor cell of the surgical specimen.

Since radiotherapy has been proven to help reduce local recurrence and improve survival rate as postoperative adjuvant treatment in patients who have undergone Breast-Conserving Surgery, a study in Nipple-Sparing Mastectomy also has been conducted to reduce local recurrence.

Benediksson's research team have reported, radiotherapy reduced the local recurrence rate in patients who had undergone Nipple-Sparing Mastectomy with reconstruction.

Petit's research team reported, the local recurrence rate is 1.7% and there was no recurrence near Nipple-Areola Complex in patients who received Nipple-Sparing Mastectomy.

Among the 486 patients who have undergone Nipple-Sparing Mastectomy with reconstruction from January 2012 to December 2017 in National Cancer Center in Korea, the local recurrence rate is 8.2%, 5% of the nipple-areola complex, 2.2% of axillary lymph node, 0.9% of the chest wall. And most of the local recurrence sites were nipple-areola complex and axillary lymph node.

Despite reducing recurrence rate, as an influencing factor to postoperative complications and cosmetics, radiotherapy has a risk of side effects from the Nipple-Sparing Mastectomy with reconstruction-operated patients.

Therefore, by conducting a prospective observational study of radiation therapy to the nipple-areola complex(close resection margin at primary tumor site) or regional lymph nodes(including axilla and supraclavicular lymph node) with a high risk of local recurrence in nipple-sparing mastectomy with reconstruction, we're going to analysis the effects of radiation therapy and cosmetic effects.

By evaluating survival rate, recurrence pattern(local lymph node and metastasis to the whole body), side effects, cosmetic effects, from the patients who have gone through Nipple Sparing Mastectomy with reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. patient who have pathologic confirmation of Ductal carcinoma in situ or invasive caricinoma
2. patient who undergone nipple sparing mastectomy with construction
3. patient who considered radiotherapy in breast cancer at stage IIB or lower (exclude ≥T3, ≥N2)
4. patient who have not distant metastasis
5. age >19 years old
6. patinet who have an ECOG of 0-2
7. patient who have not comorbidities(collagne vascular disease, such as systemic lupus erythermatosis, scleroderma, dermatomyositis)
8. patient who have not prior radiotherapy history in treatment site
9. patient who have not pregnancy or lacting
10. patient who have consent in writing to participate in research

Exclusion Criteria:

1. patient who undergone construction after nipple sparing mastectomy
2. patient who have ≥T3, ≥N2 in breast cancer
3. patient who have diastant metastasis
4. patient who have comorbidities(collagne vascular disease, such as systemic lupus erythermatosis, scleroderma, dermatomyositis)
5. patient who have treatment history in treatment site
6. patinet who have an ECOG 3-4
7. age < 20years old
8. patient who have pregnancy or lacting
9. patient who have not consent in writing to participate in research

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients receiving nipple sparing mastectomy with breast reconstruction
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
freedom from local and regioanl recurrence rate : FFLRR rate | up to 5 years
  evaluate the freedom from local and regioanl recurrence rate in nipple-areola complex(close resection margin at primary tumor site) or regional lymph nodes(including axilla and supraclavicular lymph node)

SECONDARY OUTCOMES:
relapse-free or overall survivor : RFS and OS | up to 5 years
  evaluate the Relapse-free or overall survivor in nipple-areola complex(close resection margin at primary tumor site) or regional lymph nodes(including axilla and supraclavicular lymph node)
toxicity and contraction of the implant, quality of life | up to 5 years
  evaluate the toxicity about breast site, implant surgical complication and contraction, hematopoietic.
  The quality of life is evaluated with the questionnaire filled out by the study subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tae hyun Kim, Ph.D, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea